CLINICAL TRIAL: NCT00149006
Title: Tumor-Selective and Systemic Cell Therapy of Cancer With Allogeneic Blood Lymphocytes Activated With rIL-2 and Non-Myeloablative Stem Cell Transplantation
Brief Title: Cell Therapy of Cancer With Allogeneic Blood Lymphocytes Activated With Recombinant Interleukin-2 (rIL-2) for Metastatic Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 271296-HMO-CTIL
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2007-03-14 (Estimated); Status verified 2005-09

CONDITIONS: Tumors
Keywords: Metastatic solid tumor; Mismatch allogeneic cell mediated immunotherapy
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Cell- and Tissue-Based Therapy

INTERVENTIONS:
Procedure: Cell therapy

SUMMARY:
The present protocol is designed to investigate the potential application of allogeneic cell-mediated immunotherapy in metastatic solid tumors similarly to the well established graft versus leukemia (GVL) effects in patients with hematologic malignancies.

Patients with metastatic solid tumors resistant to conventional modalities will be eligible to participate in a treatment program based on the administration of non-myeloablative immunotherapy (i.e. fludarabine, Cytoxan) followed by interferon injections; subsequently the patients will be treated with mismatched alloreactive donor lymphocytes activated in vitro and in vivo with rIL-2. The aim of this study is based on the recognition of foreign tumor cell surface alloantigens.

ELIGIBILITY:
Inclusion Criteria:

Consenting patients (age < 70) will be eligible for participation in the study involving selective anti-tumor immunotherapy provided the following criteria are met:

* Evidence of cancer not expected to be cured with conventional modalities
* Pediatric patients: Chemotherapy-resistant neuroblastoma stage 4 and sarcomas. Adult patients: Metastatic breast cancer, malignant melanoma, renal cell cancer and selected cases of ovarian cancer, gastrointestinal cancer, small-cell and non-small cell lung cancer with non-bulky metastatic disease, and metastatic prostate cancer.
* Patients with measurable disease evaluable for response with anticipated life expectancy > 3 months.
* Patients must be > 2 weeks off of anti-cancer or potentially immunosuppressive treatment.
* Adequate ambulatory performance status (Karnofsky > 80%; ECOG 0-1) to enable outpatient treatment.
* Compliant and cooperative patients anticipated to be evaluable for response according to the investigator's assessment.
* HLA-compatible (fully matched or single locus mismatched) donor available for allogeneic stem cell transplantation.

Exclusion Criteria:

* Patients with bulky disease or patients with brain metastases resistant to chemo-radiotherapy.
* Patients with a significant history or current evidence of potentially severe cardiovascular or lung disease, or other disease or clinical condition that may not permit accomplishing the planned treatment or drawing conclusions.
* Hepatic and/or renal failure.
* Evidence of serious active infection requiring antibiotic therapy.
* Pregnancy.
* Contraindication for donation due to donor disease: HIV-1; hepatitis B surface antigen (HBsAg) positivity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 1996-12

PRIMARY OUTCOMES:
Study the feasibility, toxicity, and response rate of allogeneic cell therapy induced by selective intra-lesional and systemic administration of mismatched alloreactive lymphocytes in patients with metastatic cancer

SECONDARY OUTCOMES:
Study the feasibility, toxicity, and response to treatment with allogeneic mini-transplant using sibling donors in patients with metastatic cancer

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Slavin, MD, Principal Investigator — Hadassah Medical Organization; Reuven Or, MD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel